CLINICAL TRIAL: NCT05819775
Title: A Phase 3 Open-label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of CSL312 (Garadacimab) in the Prophylactic Treatment of Hereditary Angioedema in Pediatric Subjects 2 to 11 Years of Age
Brief Title: CSL312_3003 Safety and Pharmacokinetic Study in Subjects 2 to 11 Years of Age With Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL312_3003; 2022-502386-13-00 (EU CTIS Number)
Record Dates: First submitted 2023-04-04; First posted 2023-04-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CSL312 (Experimental): Ages 2-5 years and 6-11 years will have specific subcutaneous dosing schedules
  Interventions: Biological: CSL312

INTERVENTIONS:
Biological: CSL312 — Fully human immunoglobulin G subclass 4/lambda recombinant inhibitor monoclonal antibody administered subcutaneously (SC)
  Other Names: Garadacimab

SUMMARY:
The purpose of this study is to investigate the safety, PK / PD, and efficacy of SC CSL312 for prophylactic treatment of pediatric subjects with HAE.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female
* 2. Aged 2 to 11 years, inclusive, with body weight ? 10th percentile based on age
* 3. Diagnosed with clinically confirmed C1-INH HAE
* 4. Experienced ? 2 HAE attacks during the 6 months before Screening

Exclusion Criteria:

* 1. Concomitant diagnosis of another form of angioedema, such as idiopathic or acquired angioedema, recurrent angioedema associated with urticaria, or HAE type 3
* 2. Use of C1-INH products, androgens, antifibrinolytics, approved or future approved medications, or other small molecule medications for routine prophylaxis against HAE attacks within a minimum of 2 weeks before the Treatment Period
* 3. Participation in another interventional clinical study during the 30 days before the Treatment Period or within 5 half-lives of the final dose of the investigational product administered during the previous interventional study, whichever is longer
* 4. Having laboratory clinical abnormalities assessed as clinically significant by the investigator in results of hematology or chemistry assessments performed during Screening
* 5. Currently receiving a therapy not permitted during the study
* 6. Being pregnant or breastfeeding.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) | At least 14 months
Percent of subjects with TEAEs | At lease 14 months
Number of TEAEs | At least 14 months
TEAE rates per injection | At least 14 months
TEAE rates per subject year | At least 14 months
Maximum concentration (Cmax) of CSL312 at steady-state | At least 12 months
Trough concentration (Ctrough) of CSL312 at steady-state | At least 12 months
Time to maximum concentration (Tmax) of CSL312 at steady-state | At least 12 months

SECONDARY OUTCOMES:
Time-normalized number of HAE attacks per month and per year | At least 12 months
Time-normalized number of HAE attacks treated with on-demand treatment per month and per year | At least 12 months
Time-normalized number of moderate and / or severe HAE attacks per month and per year | At least 12 months
Percentage reduction in the time-normalized number of HAE attacks | At least 12 months
The number of subjects experiencing at least ? 50%, ? 70%, ? 90%, or equal to 100% (attack-free) reduction in the time-normalized number of HAE attacks | At least 12 months
Number of subjects with serious adverse events (SAEs) | At least 14 months
Percent of subjects with SAEs | At least 14 months
Number of subjects experiencing death | At least 14 months
Percent of subjects experiencing death | At least 14 months
Number of subjects with related TEAEs | At least 14 months
Percent of subjects with related TEAEs | At least 14 months
Number of subjects with TEAEs leading to study discontinuation | At least 14 months
Percent of subjects with TEAEs leading to study discontinuation | At least 14 months
Number of subjects with TEAEs by severity | At least 14 months
Percent of subjects with TEAEs by severity | At least 14 months
Number of subjects with Anti-CSL312 antibodies | At least 14 months
Percent of subjects with Anti-CSL312 antibodies | At least 14 months
Number of subjects with adverse events of special interest (AESIs) | At least 14 months
Percent of subjects with AESIs | At least 14 months
FXIIa-mediated kallikrein activity | At least 12 months
  Blood samples will be collected on the same day as CSL312 administration for assessment of FXIIa-mediated kallikrein activity
Number of subjects with laboratory findings reported as AEs | At least 14 months
Percent of subjects with laboratory findings reported as AEs | At least 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (13):
- United States (7):
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Medical Research of Arizona, Scottsdale, Arizona
  - Donald S. Levy M.D., Orange, California
  - Raffi Tachdjian MD, Inc., Santa Monica, California
  - Bernstein Clinical Research, Cincinnati, Ohio
  - PennState Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Campbelltown Hospital, Western Sydney University, Campbelltown, Australia
- Ottawa Allergy Research Corp, Ottawa, Canada
- Germany (3):
  - HZRM Hämophilie Zentrum Rhein Main GmbH, Frankfurt am Main, Hesse
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
- Barzilai University Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.